CLINICAL TRIAL: NCT05917821
Title: Identification of New Antigens Against Glioblastoma
Brief Title: New Antigens Against Glioblastoma
Acronym: INAAG
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5866
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators will select and develop potential therapeutic monoclonal antibodies (mAbs) for glioblastoma (GB). Activities include tissue microarray (TMA) to test monoclonal antibodies specificity and target distribution, selection of glioblastoma specific functional monoclonal antibodies, identification of candidate targets.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* Written informed consent

Exclusion Criteria:

* Not-availability of informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: National monocentric study, enrolling approximately 120 patients with glioblastoma, males and females, no pedriatic age.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Validation of the tumour specificity of the identified monoclonal antibodies | 4 years
  Candidate monoclonal antibodies will be tested by immunohistochemistry (IHC) on sections of glioblastoma tissue and healthy counterpart.

SECONDARY OUTCOMES:
Generate the single chain Fab antibody fragments (scFv) and then develop the Chimeric Antigen Receptor (CAR) T cells | 4 years
  After defining a subset of potentially highly selective ~7 monoclonal antibodies, together with the ~6 that showed preliminary activity in cytotoxic tests (either alone or conjugated), the investigators will perform a thorough analysis of their specificity on a TMA platform. After establishing the staining conditions, the investigators will test multiple tumor and multiple normal TMAs